CLINICAL TRIAL: NCT00740350
Title: Does the Logan Basic Protocol for Chiropractic Care During Pregnancy Reduce Labor Time and Increase the Ease of Labor and Childbirth?
Brief Title: Logan Basic During Pregnancy on Labor and Childbirth
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Patrick Montgomery, DC, Logan University, College of Chiropractic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SR0627080139
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Logan Basic chiropractic adjustments during pregnancy.
  Interventions: Procedure: Logan Basic

INTERVENTIONS:
Procedure: Logan Basic — Logan Basic chiropractic adjustments during pregnancy.

SUMMARY:
The purpose of this study is to determine if women who have chiropractic care, according to the Logan Basic Protocol for adjusting, during pregnancy have an easier, shorter labor and delivery as compared to women who haven't had chiropractic care during pregnancy.

DETAILED DESCRIPTION:
This study will be designed to test if the Logan Basic Technique system of adjusting pregnant women can reduce labor time and increase the ease of labor and delivery as compared to the labor times reported by Kilpatrick and Laros in the obstetric literature. It is proposed that women who have regular chiropractic care throughout pregnancy or at least for the third trimester will have an easier labor and delivery as well as a shorter labor time than is reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* 20-24 weeks pregnant
* enrolled in a separate pre-natal care protocol with an outside provider
* a Logan College Student or member of the family of a Logan Student ("family" as defined by CCE designation)

Exclusion Criteria:

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Post delivery interview/questionnaire | 2 weeks post delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States